CLINICAL TRIAL: NCT06205602
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Combination of Two Long-Acting Broadly Neutralizing Antibodies at ART Initiation in Adults Living With HIV-1 in Sub-Saharan Africa: The ACACIA Study
Brief Title: Antiretrovirals Combined With Antibodies for HIV-1 Cure In Africa
Acronym: ACACIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5417; UM1AI068636 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Broadly neutralizing antibodies (bNAbs) infusions with antiretroviral therapy (ART) (Active Comparator)
  Interventions: Drug: 3BNC117-LS; Drug: 10-1074-LS
- Placebo infusions with ART (Placebo Comparator)
  Interventions: Drug: Placebo for 3BNC117-LS; Drug: Placebo for 10-1074-LS

INTERVENTIONS:
Drug: 3BNC117-LS — 30 mg/kg to be administered via IV at Step 1 (Day 1)
  Arms: Broadly neutralizing antibodies (bNAbs) infusions with antiretroviral therapy (ART)
Drug: 10-1074-LS — 10 mg/kg to be administered intravenously at Step 1 (Day 1)
  Arms: Broadly neutralizing antibodies (bNAbs) infusions with antiretroviral therapy (ART)
Drug: Placebo for 3BNC117-LS — 0.9% Sodium Chloride Injection to be administered intravenously at Step 1 (Day 1)
  Arms: Placebo infusions with ART
Drug: Placebo for 10-1074-LS — 0.9% Sodium Chloride Injection) to be administered IV at Step 1 (Day 1)
  Arms: Placebo infusions with ART

SUMMARY:
For people living with HIV, antiretroviral therapy (ART) helps to stop the virus from multiplying. The goal of current HIV treatment is to have such a small amount of the virus in the blood that it does not show up on regular tests. HIV is also hidden in cells throughout the body and can start multiplying when ART is stopped.

This research study will test two new study drugs: 10-1074-LS and 3BNC117-LS. Both of these study drugs are antibodies against HIV. An antibody is generally a substance that the body makes in response to an infection. The antibodies being used in this study were made in a laboratory and were designed to attach to HIV and can block HIV from attacking cells in the body and from spreading to other parts of the body. These antibodies are being developed to potentially treat and prevent HIV.

The main purpose of this study is to see if the study drugs affect the level of HIV that remains in the blood cells while taking ART and the level of HIV in the blood after discontinuing taking ART. The study will also see if it is safe to give people these antibodies and if they cause any side effects.

ELIGIBILITY:
Step 1 Inclusion Criteria:

* Confirmed HIV-1, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study Step 1 entry AND Confirmed by one of the following:

  * A second antibody test from different manufacturers or based on different principles and epitopes (combination antigen-antibody-based rapid tests may be used)
  * HIV-1 antigen
  * Plasma HIV-1 RNA viral load or
  * A licensed Western blot

NOTE: The term "licensed" refers to a US FDA or DAIDS Clinical Laboratory Oversight (DCLOT) approved test.

WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

* ART-naïve [NOTE: Prior use of PrEP or PEP is allowed, except use of long-acting ARVs (e.g., cabotegravir, rilpivirine) within the last 24 months.]
* CD4+ T cell count >200 cells/mm3 obtained within 28 days prior to study entry at any Network-approved non-US laboratory that is (IQA) certified.
* Plasma HIV-1 RNA >1000 copies/mL obtained within 28 days prior to study entry performed at any Network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate external quality assurance (EQA) programs.
* For study candidates of child-bearing potential, negative urine or serum pregnancy test within 72 hours prior to study entry by any Network-approved non-US laboratory or clinic that operates in accordance with GCLP and participates in appropriate EQA programs.

[NOTE A: Persons who are of child-bearing potential are individuals who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, and who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy, tubal ligation, or bilateral salpingectomy.] [NOTE B: Acceptable documentation of hysterectomy and bilateral oophorectomy, tubal ligation, and tubal micro-inserts are written documentation or oral communication from a clinician or clinician's staff documented in source documents (physician report/letter, operative report or other source documentation in the patient record, discharge summary, laboratory report, etc.). Participant-reported history is acceptable for documentation of menopause.]

* Persons of child-bearing potential who are able to become pregnant must agree to use two methods of contraception, if participating in sexual activity that could lead to pregnancy. One contraceptive method must be from the list of highly effective methods listed below. The second method of contraception must be a barrier method or abstinence. Both methods of contraception must be used during Step 1. The two effective forms of birth control have to be used for 10 days before receiving the first study drug infusion, for at least 12 months after the product infusion, and until ART is reinitiated and viral suppression is achieved.

Acceptable methods of contraception include:

* Contraceptive subdermal implant
* Intrauterine device or intrauterine system
* Combined estrogen and progestogen oral contraceptive
* Injectable progestogen
* Contraceptive vaginal ring
* Percutaneous contraceptive patches
* Partner sterilization with documentation of azoospermia prior to the participant's entry into the study, and this individual is the sole partner for that participant.

[NOTE: Documentation of partner sterility can come from the site personnel's review of participant's medical records, medical examination and/or semen analysis, or medical history interview provided by the participant or the partner. Self-reported documentation of reproductive potential should be entered in the source documents.]

* Individuals engaging in sexual activity that could lead to their partner becoming pregnant must agree to use a barrier method of contraception to avoid pregnancy in a spouse or partner of reproductive potential. The barrier method must be used to prevent partner pregnancy during Step 1 and for at least 12 months after the product infusion.
* Ability and willingness to use a barrier protection or abstinence from sexual intercourse during Step 1 until viral suppression is achieved, during the ATI period (Steps 2-3), and until plasma HIV-1 RNA is less than limit of detection after ART restart (Step 4) with partners without HIV or whose HIV serostatus is unknown in order to prevent HIV transmission to sexual partners.
* Ability and willingness to initiate ART at enrollment.
* Ability and willingness to participate in scheduled study visits, including ATI per the SOE.
* Ability and willingness to provide informed consent.

Step 2 Inclusion Criteria:

* Documented negative hepatitis B virus (HBV) surface antigen (HBsAg) obtained within 16 weeks prior to Step 2 registration by any Network-approved non-US laboratory that operates in accordance with GCLP and participates in appropriate EQA programs.
* Documented negative HCV antibody (anti-HCV), negative HCV RNA PCR, or negative HCV antigen obtained within 16 weeks prior to Step 2 registration by any Network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate EQA programs.
* Participants diagnosed with a bacterial sexually transmitted infection (STI) must have initiated treatment prior to Step 2 entry.
* Receipt of both bNAb infusions or placebo infusions during Step 1.
* HIV-1 RNA <200 copies/mL obtained within 6 weeks prior to Step 2 registration at any Network-approved non-US laboratory that is VQA certified.
* CD4+ T cell count ≥450 cells/mm3 obtained within 6 weeks prior to Step 2 registration at any Network-approved non-US laboratory that is IQA certified.
* For participants of child-bearing potential, negative serum or urine pregnancy test within 48 hours prior to Step 2 entry at any Network-approved non-US laboratory or clinic that operates in accordance with GCLP and participates in appropriate EQA programs.
* Ability and willingness to use a barrier method of contraception or abstinence from sexual intercourse during Steps 2 and 3, and until plasma HIV-1 RNA is less than limit of detection, with all partners who are without HIV or whose serostatus is unknown in order to prevent HIV transmission to sexual partners.
* Ability and willingness to stop ART.

Step 3 Inclusion Criteria

* Has not met ART restart criteria.
* Completion of protocol Step 2.
* Willing to continue ATI.

Step 4 Inclusion Criteria

* Met ART restart criteria (section 3.0) during Step 2 or Step 3 OR Completed Step 3 and is not enrolling to ACTG A5385.

Step 1 Exclusion Criteria:

* Any clinically significant acute or chronic medical condition, other than HIV, that in the opinion of the investigator would preclude safe participation in the study or interfere with the validity of study results.
* Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months. [NOTE: Minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) are not exclusionary.]
* History of AIDS-defining illness within 3 years prior to enrollment.
* History of systemic corticosteroids (e.g., an equivalent dose of prednisone of > 20 mg daily for >14 days), immunosuppressive anti-cancer, interleukins, systemic interferons, systemic chemotherapy or other medications considered significant by the trial physician within the last 12 weeks.
* History of a severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis in the 2 years prior to enrollment.
* History of chronic urticaria requiring current daily treatment.
* Known history of active Hepatitis B or Hepatitis C infection. [NOTE: Participant is eligible if hepatitis C virus (HCV) cure or clearance is documented.]
* History of or current clinical atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 American College of Cardiology (ACC)/American Heart Association (AHA) guidelines, including a previous diagnosis of any of the following:

  * Acute myocardial infarction
  * Acute coronary syndromes
  * Stable or unstable angina
  * Coronary or other arterial revascularization
  * Stroke
  * Transient ischemic attack
  * Peripheral arterial disease presumed to be of atherosclerotic origin
* Any history of receipt of HIV vaccine candidate or HIV-specific monoclonal antibody therapy.
* Participation in any clinical study of an investigational product within 28 days prior to study entry (day 0) or expected participation in such a study during participation in this study. [NOTE: Treatment or receipt of prophylaxis against other infectious pathogens such as SARS-CoV-2 or Monkeypox under Emergency Use Authorization within 28 days of study entry is not exclusionary.]
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Breastfeeding
* Laboratory abnormalities in the parameters listed below, obtained by any Network-approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practices (GCLP) and participates in appropriate EQA programs.

  * Absolute neutrophil count <750 cells/mm3
  * Hemoglobin <9 gm/dL for volunteers who were assigned female sex at birth, <10.0 g/dL for volunteers who were assigned male sex at birth
  * Platelet count <100,000 cells/mm3
  * ALT >3 x ULN
  * AST >3 x ULN
  * Total bilirubin >2 x ULN
  * eGFR <60 mL/min/1.73m2
* Use of prohibited medications with ART within 7 days prior to study entry, or planned use of prohibited medications during the period of study participation.

[NOTE: Use of St. John's wort within 7 days prior to study entry is acceptable but must be discontinued on the day of study entry]

Step 2 Exclusion Criteria:

* Viral failure after Step 1 week 24.
* Participant never started ART.
* Participant interrupted ART ≥7 consecutive days in Step 1.
* Current use of an ART regimen that includes a long-acting or NNRTI component.
* Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during ATI.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Step 3 Exclusion Criteria

* Transfer to A5385 (The Post-Intervention Cohort Study) [NOTE: Participants may be offered co-enrollment or transfer to A5385, depending on ACTG identification of the preferred methodology for observation during extended ATI.]
* Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during analytic treatment interruption.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Step 4 Exclusion Criteria

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2029-02-16 (Estimated); Study Completion 2029-02-16 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade ≥2 Adverse Events (AE) or Serious Adverse Events (SAE) | Day 0 through Week 56
  Occurrence of Grade ≥2 AE or SAE that are possibly, probably, or definitely related to the study bNAbs during Step 1 (as judged by the CMC, blinded to active/placebo treatment).
Time from antiretroviral therapy (ART) discontinuation to sustained HIV-1 RNA ≥ 1000 copies/mL over a 4-week period (through step 2) | 4 weeks from Step 2 Day 0 (Study week 60, 72 or 84 depending on early pharmacokinetic modeling)
  Sustained HIV-1 RNA ≥1000 copies/mL over a 4-week period means at least two measurements of HIV-1 RNA ≥1000 copies/mL over 4 weeks with no HIV-1 RNA <1000 copies/mL measured between them. Through Step 2 means the 4-week period has started between Step 2 week 0 and week 24.Time to sustained HIV-1 RNA ≥1000 copies/mL over 4 weeks is the time to the first measurement that reaches that level over 4 weeks.

SECONDARY OUTCOMES:
Time from ART discontinuation to ART restart | Time from ART discontinuation (can occur at 60, 72 or 84 weeks) to restart of ART (0 to 72 weeks after ART discontinuation)
  Time between ART discontinuation to the time participant meeting virologic, immunologic or clinical criteria (i.e., viral load, CD4+ T cell count, or development of severe acute retroviral syndrome) for ART restart
The proportion of participants who undergo ATI without indication of ART restart | Time from ART interruption(study week 60, 72 or 84) through 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Crowell, MD, PhD, Study Chair — US Military HIV Research Program CTU; Wadzanai Samaneka, MBChB, MSc, Study Chair — Milton Park CRS
Locations (4):
- Gaborone CRS (12701), Gaborone, Botswana
- South Africa (3):
  - University of the Witwatersrand Helen Joseph (WITS HJH) CRS (11101), Johannesburg, Gauteng
  - CAPRISA eThekwini CRS (31422), Durban, KwaZulu-Natal
  - Durban Adult HIV CRS (11201), Durban

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
  Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at:
  https://actgnetwork.org/submit-a-proposal-2/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.